CLINICAL TRIAL: NCT02023203
Title: Prospective Randomized Clinical Trial Comparing Microporous Polypropylene Mesh and Flexible Macroporous Polytetrafluoroethylene Mesh in Totally Extraperitoneal Laparoscopic Inguinal Hernia Repair
Brief Title: Efficacy of Macroporous Polytetrafluoroethylene Mesh in Laparoscopic Hernia Repair
Acronym: PTFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Principal Investigator, Salvador Morales Conde, Innovation and Minimally Invasive Surgery Unit Cordinator, Hospitales Universitarios Virgen del Rocío
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LP-PTFE
Record Dates: First submitted 2013-12-13; First posted 2013-12-30 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Hernia, Inguinal
MeSH Terms: conditions — Hernia, Inguinal | interventions — tetraethylpyrazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LP PTFE (Experimental): Placement of Large Pore PTFE mesh for inguinal hernia treatment
  Interventions: Procedure: Totally Extraperitoneal laparoscopic inguinal hernia repair
- SP-PPL (Active Comparator): Placement of Small Pore polypropylene mesh for inguinal hernia treatment
  Interventions: Procedure: Totally Extraperitoneal laparoscopic inguinal hernia repair

INTERVENTIONS:
Procedure: Totally Extraperitoneal laparoscopic inguinal hernia repair — Laparoscopic hernioplasty
  Other Names: TEP

SUMMARY:
Inguinal hernia repair is one of the most commonly performed surgeries around the world. It accounts for approximately 75% of all abdominal wall hernias and presents a lifetime risk of 27% in males and 3% in females. Since the modern concept of surgical hernia repair described by Bassini in 1887, with the technique that bears his name, several techniques have been developed in the last century in order to improve surgical outcomes after inguinal hernia repair.

Different open repairs, such as anterior (Shouldice, McVay) or posterior (Stoppa) approach were described and developed, until Lichtenstein described the tension-free hernioplasty concept supported by the use of a prosthetic mesh to repair the hernia defect. Notable Improvements were observed with this technique in terms of recurrence, pain, and discomfort in comparison with previous tension repairs. Considerable advantages over open repair have been obtained with the introduction of minimally invasive surgery to inguinal hernia repair, in terms of patient comfort and recurrence rates.

Regarding prosthetic material, meshes have evolved since the first Dacron mesh used by Lichtenstein. First generation meshes were manufactured using more material and for this reason they have been described as heavyweight meshes. New generation meshes have been designed with less material in order to diminish the inflammatory response and foreign body reaction, providing less chronic pain with similar recurrence rates than heavyweight meshes. The density (or weight) of the mesh, measured in g/m2, is inversely proportional to the size of the pore and lately it has been reported that one of the main aspects related to prosthetic materials is pore size. Large pore meshes use less material, consequently they have been associated with a better tissue ingrowth. The large pore of lightweight meshes is conditioned by the less amount of material used.

All previous studies compare both light and heavyweight polypropylene meshes But in order to get a proper comparison of the behavior of meshes in the inguinal region it is important to include the material and the pore size. The aim of our study is to compare patient-reported outcomes with the use of either a Polytetrafluoroethylene (PTFE) large pore mesh (LP-PTFE) vs a small pore polypropylene mesh (SP-PPL).

DETAILED DESCRIPTION:
Patients fitted for laparoscopic bilateral inguinal hernia repair will be randomized to recieve one of both meshes on study in both inguinal sides.

ELIGIBILITY:
Inclusion Criteria:

* male patients
* 20-80 years old
* Primary Bilateral Hernia

Exclusion Criteria:

* Women
* BMI >35
* Recurrent hernias
* Previous infraumbilical laparotomy
* Inguinoscrotal hernias

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2012-10 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Postoperative Discomfort | 1 year
  Postoperative Discomfort in the inguinal area is assessed using a visual analog scale (VAS)on the first 12 postoperative months.
  Discomfort is defined as a disturbing sensation without influencing normal activities of the patient

SECONDARY OUTCOMES:
Postoperative Pain | 1 year
  Postoperative pain in the inguinal area is assessed using a visual analog scale (VAS)on the first 12 postoperative months.
  Pain is described as an unpleasant sensation that interferes with the normal activities of the patient
Recurrence | 1 year
  Reappearance of a inguinal hernia in a previous operated inguinal hernia.
Postoperative complications | 1 year
  Complications such as seroma or haematoma in groin area.

CONTACTS AND LOCATIONS:
Overall Officials: Salvador Morales-Conde, PhD, Principal Investigator — Hospital Universitario Virgen del Rocio; Isaias Alarcón, PhD, Study Chair — Hospital Universitario Virgen del Rocio
Locations (1):
- Hospital Universitario Virgen del Rocio, Seville, Seville, Spain

REFERENCES:
- [Background] Pascual G, Hernandez-Gascon B, Rodriguez M, Sotomayor S, Pena E, Calvo B, Bellon JM. The long-term behavior of lightweight and heavyweight meshes used to repair abdominal wall defects is determined by the host tissue repair process provoked by the mesh. Surgery. 2012 Nov;152(5):886-95. doi: 10.1016/j.surg.2012.03.009. Epub 2012 May 8. PMID 22575883
- [Background] Jacob DA, Schug-Pass C, Sommerer F, Tannapfel A, Lippert H, Kockerling F. Comparison of a lightweight polypropylene mesh (Optilene(R) LP) and a large-pore knitted PTFE mesh (GORE(R) INFINIT(R) mesh)--Biocompatibility in a standardized endoscopic extraperitoneal hernia model. Langenbecks Arch Surg. 2012 Feb;397(2):283-9. doi: 10.1007/s00423-011-0858-8. Epub 2011 Oct 12. PMID 21989559
- [Background] Melman L, Jenkins ED, Hamilton NA, Bender LC, Brodt MD, Deeken CR, Greco SC, Frisella MM, Matthews BD. Histologic and biomechanical evaluation of a novel macroporous polytetrafluoroethylene knit mesh compared to lightweight and heavyweight polypropylene mesh in a porcine model of ventral incisional hernia repair. Hernia. 2011 Aug;15(4):423-31. doi: 10.1007/s10029-011-0787-z. Epub 2011 Jan 30. PMID 21279663
- [Derived] Alarcon I, Balla A, Soler Frias JR, Barranco A, Bellido Luque J, Morales-Conde S. Polytetrafluoroethylene versus polypropylene mesh during laparoscopic totally extraperitoneal (TEP) repair of inguinal hernia: short- and long-term results of a double-blind clinical randomized controlled trial. Hernia. 2020 Oct;24(5):1011-1018. doi: 10.1007/s10029-020-02200-y. Epub 2020 Apr 30. PMID 32350735